CLINICAL TRIAL: NCT05577897
Title: The Effects of Education Given to Patients Diagnosed With Chronic Obstructive Pulmonary Disease on Self-care Agency and Rational Drug Use.
Brief Title: Effectiveness of Education Given to Patients With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeynep Yildirim (Other)
Responsible Party: Sponsor-Investigator, Zeynep Yildirim, Research Assistant, Ataturk University
Organization: Ataturk University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Zeynep
Record Dates: First submitted 2022-09-27; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: COPD
Keywords: Patient education; Nurse; COPD; Self-care agency; Rational drug use
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Education (Experimental): The intervention group was given 45 minutes of training.
  Interventions: Other: Education
- Control Group (No Intervention): Routine nursing care was given to the patients in this group without any training.

INTERVENTIONS:
Other: Education — A separate room in Chest Diseases Clinic was used for the education of the patients in this group for a quiet environment and for the education not to be interrupted. The education of a patient lasted approximately 45 minutes. The education booklet "COPD Guide" on COPD management prepared in line with the literature was given to the patients by the researcher. After the content of the education was explained to the patients, 45-minute of education was given through face-to-face verbal presentation and demonstration method.
  Arms: Patient Education

SUMMARY:
This study was conducted to examine the effects of chronic obstructive pulmonary disease management education given to patients diagnosed with chronic obstructive pulmonary disease on self-care agency and rational drug use. This study has a pretest-posttest quasi-experimental design. A total of 83 patients with COPD were randomly assigned to a intervention group or control group, who met the inclusion criteria.

DETAILED DESCRIPTION:
COPD, which is one of the most common respiratory system diseases, is an important global health problem. Chronic Obstructive Pulmonary Disease (COPD), which is a disease with significant mortality and morbidity, is characterized by progressive air flow obstruction; it is irreversible and accompanied by multiple symptoms and frequent exacerbations. Among the leading causes of death, COPD is in the fourth place in the world, while it is in the third place in our country.

At the end of the physiopathological processes that occur in COPD, respiratory function is severely impaired, and individuals experience significant levels of limitations while performing their daily living activities due to shortness of breath, cough, fatigue and insomnia. Long-term drug therapy is used commonly to control these limitations in patients with COPD. Increased dyspnea, activity intolerance, long lasting oxygen and drug therapy, social intolerance and chronic hypoxia cause a decrease in the quality of life and psychological problems. It is important for patients to have sufficient level of self-care agency and to take responsibility for their self-care to control COPD symptoms. Self-care management consists of behaviors performed to manage the symptoms of the disease or to manage the side effects of the treatment. In patients with COPD, self-care is specifically important since it can improve health-related quality of life and decrease hospitalization and dispnea.

One of the necessary steps to improve the symptoms and limitations caused by the physiopathological processes that occur in COPD is drug therapy. A large number of drug groups are used in COPD treatment. The aim of drug therapy in COPD is eliminating the symptoms, improving exercise tolerance and health status and increasing future risks (prevention and treatment of attacks, prevention of disease progression and decrease in mortality). Stable COPD treatment should be individualized depending on the symptoms of patients. In patients with COPD, the problem of compliance with medication due to reasons such as insufficient or no training on medication, cognitive or physical insufficiency of patients, educational and sociocultural level difference of patients, not choosing the device suitable for patients, misuse of drug, or the inability to use the drug are very common among patients. Patients should be able to transform rational drug use into behavior and have the required knowledge and attitude levels. In this context, the responsibility of nurses for educating and informing patients emerges.

Education is very important in terms of improving the self-care skills of patients with COPD, increasing their functional abilities, using drugs properly, managing the disease processes and improving quality of life. The effects of the education given on different parameters have been evaluated in literature. Therefore, it is thought that the education given to patients about COPD management may contribute to increasing the self-care agency of the patient and to rational use of drugs. This study was conducted to find out the effects of COPD management education given to patients diagnosed with COPD on self-care agency and rational drug use.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had been receiving CODP treatment for longer than 6 months
* Patients who had low or moderate levels of self-care agency
* Patients who needed to use medication continuously to treat COPD
* Patients who had no sensory loss related to hearing and vision
* Patients who were open to cooperation and communication and who were oriented

Exclusion Criteria:

* Patients who left the study at any stage
* Patients who had been receiving CODP treatment for less than 6 months

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2020-12-11 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2021-07-12 (Actual)

PRIMARY OUTCOMES:
Self Care Agency Scale | up to 6 weeks
  SCAS was developed by Kearney and Fleischer. It was adapted into Turkish by by Nahcivan on healthy young individuals and by Pınar on chronic diseases. SCAS has 35 questions with answers on a 5-point, Likert-type scale (from 1 to 5). A total score below 82 is evaluated as low level of self-care agency, while total score between 82 and 120 is evaluated as moderate level of self-care agency and a total score higher than 120 is evaluated as high level of self-care agency.
Rational Drug Use Scale | up to 6 weeks
  RDUS was developed by Demirtaş et al. to determine rational drug use knowledge levels of adult patients. The 3 Likert-type scale consists of a total of 21 expressions, 10 correct and 11 incorrect. The answers given; Correct answer is scored as 2, I don't know 1, and wrong answer is 0 points. Maximum possible score of the scale is 42. A total score of 35 and higher is evaluated as having rational drug use knowledge.

CONTACTS AND LOCATIONS:
Locations (1):
- Zeynep YILDIRIM, Erzurum, Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No